CLINICAL TRIAL: NCT03769090
Title: A Long-term, Randomized, Double-blind, Multicenter, Parallel-group, Phase III Study Evaluating the Efficacy and Safety of PT027 Compared to PT007 Administered as Needed in Response to Symptoms in Symptomatic Adults and Children 4 Years of Age or Older With Asthma
Brief Title: A Study to Assess the Efficacy and Safety of Budesonide/Albuterol Metered-dose Inhaler (BDA MDI/PT027) in Adults and Children 4 Years of Age or Older With Asthma
Acronym: MANDALA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bond Avillion 2 Development LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AV003
Record Dates: First submitted 2018-11-30; First posted 2018-12-07 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BDA MDI (PT027) 160/180 μg (Experimental): Budesonide/albuterol sulfate, BDA MDI, PT027 high dose
  Interventions: Combination Product: Budesonide/albuterol sulfate metered-dose inhaler 160/180 μg
- BDA MDI (PT027) 80/180 μg (Experimental): Budesonide/albuterol sulfate, BDA MDI, PT027 low dose
  Interventions: Combination Product: Budesonide/albuterol sulfate metered-dose inhaler 80/180 μg
- AS MDI (PT007) 180 µg (Active Comparator): Albuterol sulfate MDI, PT007
  Interventions: Drug: Albuterol sulfate metered-dose inhaler 180 μg

INTERVENTIONS:
Combination Product: Budesonide/albuterol sulfate metered-dose inhaler 160/180 μg — Budesonide/albuterol sulfate combination inhalation aerosol
  Arms: BDA MDI (PT027) 160/180 μg
Combination Product: Budesonide/albuterol sulfate metered-dose inhaler 80/180 μg — Budesonide/albuterol sulfate combination inhalation aerosol
  Arms: BDA MDI (PT027) 80/180 μg
Drug: Albuterol sulfate metered-dose inhaler 180 μg — Albuterol sulfate inhalation aerosol
  Arms: AS MDI (PT007) 180 µg

SUMMARY:
This is a randomized, double-blind, multicenter, parallel-group, variable-length study to compare 2 doses of BDA MDI (PT027) with AS MDI (PT007) on the time to first severe asthma exacerbation in adult, adolescent, and pediatric subjects with moderate to severe asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged ≥4 years at the time of informed consent
2. Physician diagnosis of asthma documented for at least 1 year
3. Receiving 1 of the following scheduled asthma maintenance therapies for 3 months with stable dosing for at least the last 4 weeks before Visit 1:

   * Medium-to-high-dose inhaled corticosteroid (ICS)
   * Medium-to-high-dose ICS and 1 additional maintenance therapy from the following: leukotriene receptor antagonists (LTRA), long-acting muscarinic antagonists (LAMA), or theophylline
   * Low-to-high-dose ICS in combination with long-acting β2-adrenoreceptor agonist (LABA) with or without one additional maintenance therapy from the following: LTRA, LAMA, or theophylline
4. Prebronchodilator forced expiratory volume in 1 second (FEV1) of ≥40 to <90% predicted normal value for adults and adolescents, and ≥60 to <100% predicted normal value for subjects aged 4 to 11 years after withholding specified medications including short/rapid-acting β2-adrenoreceptor agonist (SABA)
5. Demonstrate reversibility at Visit 1, with an increase in FEV1 ≥12% (and ≥200 mL for subjects aged ≥18 years) relative to baseline after administration of sponsor provided Ventolin via central spirometry. One re-test for reversibility testing is allowed within the screening period in advance of Visit 2
6. Demonstrate acceptable spirometry performance (i.e., meet American Thoracic Society/European Respiratory Society acceptability/repeatability criteria)
7. A documented history of at least 1 severe asthma exacerbation within 12 months before Visit 1
8. Able to perform acceptable and reproducible peak expiratory flow (PEF) measurements as assessed by the investigator

Exclusion Criteria:

1. Chronic obstructive pulmonary disease or other significant lung disease (e.g., chronic bronchitis, emphysema, bronchiectasis with the need of treatment, cystic fibrosis, or bronchopulmonary dysplasia)
2. Oral corticosteroid/SCS use (any dose and any indication) within 6 weeks before Visit 1
3. Chronic use of oral corticosteroids (OCS, ≥3 weeks use in 3 months prior to Visit 1)
4. Having received any marketed (e.g., omalizumab, mepolizumab, reslizumab, benralizumab) or investigational biologic within 3 months or any other prohibited medication
5. Current smokers, former smokers with >10 pack-years history, or former smokers who stopped smoking <6 months before Visit 1 (including all forms of tobacco, e-cigarettes [vaping], and marijuana)
6. Life-threatening asthma defined as any history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma related syncopal episode(s) within 5 years of Visit 1
7. Historical or current evidence of a clinically significant disease
8. Cancer not in complete remission for at least 5 years
9. Hospitalization for psychiatric disorder or attempted suicide within 1 year of Visit 1
10. History of psychiatric disease, intellectual deficiency, poor motivation, or other conditions if their magnitude is limiting informed consent validity
11. Significant abuse of alcohol or drugs

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3132 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Albers, MD, PhD, Study Director — Avillion LLP
Locations (274):
- United States (142):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Montgomery, Alabama
  - Research Site, Scottsboro, Alabama
  - Research Site, Sheffield, Alabama
  - Research Site, Tuscumbia, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Peoria, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Bakersfield, California
  - Research Site, Bellflower, California
  - Research Site, Canoga Park, California
  - Research Site, Encinitas, California
  - Research Site, Hawthorne, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Rancho Cucamonga, California
  - Research Site, Redwood City, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, San Jose, California
  - Research Site, Westminster, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Waterbury, Connecticut
  - Research Site, Aventura, Florida
  - Research Site, Boynton Beach, Florida
  - Research Site, Cape Coral, Florida
  - Research Site, Clearwater, Florida
  - Research Site, DeLand, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Greenacres City, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Oviedo, Florida
  - Research Site, Palmetto Bay, Florida
  - Research Site, Panama City, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Albany, Georgia
  - Research Site, Winder, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Normal, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Overland Park, Kansas
  - Research Site, Topeka, Kansas
  - Research Site, Owensboro, Kentucky
  - Research Site, Bangor, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Chevy Chase, Maryland
  - Research Site, White Marsh, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Fall River, Massachusetts
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Hamtramck, Michigan
  - Research Site, Rochester, Michigan
  - Research Site, Rochester Hills, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, Hazelwood, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Bellevue, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Brick, New Jersey
  - Research Site, Marlton, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Potsdam, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Monroe, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Dublin, Ohio
  - Research Site, Mayfield Heights, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Blue Bell, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Providence, Rhode Island
  - Research Site, Warwick, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Clinton, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Pelzer, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Beaumont, Texas
  - Research Site, Boerne, Texas
  - Research Site, Conroe, Texas
  - Research Site, Corsicana, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Galveston, Texas
  - Research Site, Houston, Texas
  - Research Site, Kerrville, Texas
  - Research Site, Live Oak, Texas
  - Research Site, McKinney, Texas
  - Research Site, Pearland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sherman, Texas
  - Research Site, The Woodlands, Texas
  - Research Site, Tomball, Texas
  - Research Site, Waco, Texas
  - Research Site, Waxahachie, Texas
  - Research Site, Murray, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, South Burlington, Vermont
  - Research Site, Morgantown, West Virginia
  - Research Site, Greenfield, Wisconsin
- Argentina (12):
  - Research Site, Buenos Aires
  - Research Site, Córdoba
  - Research Site, Lanús
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Quilmes
  - Research Site, Rosario
  - Research Site, Salta
  - Research Site, San Fernando
  - Research Site, San Juan Bautista
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Fe
- Canada (10):
  - Research Site, Vancouver, British Columbia
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Québec, Quebec
- Czechia (13):
  - Research Site, Beroun
  - Research Site, Brandýs nad Labem
  - Research Site, Jindřichův Hradec
  - Research Site, Kralupy nad Vltavou
  - Research Site, Kuřim
  - Research Site, Lovosice
  - Research Site, Miroslav
  - Research Site, Neratovice
  - Research Site, Prague
  - Research Site, Rokycany
  - Research Site, Tábor
  - Research Site, Teplice
  - Research Site, Varnsdorf
- Germany (34):
  - Research Site, Augsburg
  - Research Site, Bad Wörishofen
  - Research Site, Bamberg
  - Research Site, Bergisch Gladbach
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Cologne
  - Research Site, Cottbus
  - Research Site, Darmstadt
  - Research Site, Delitzsch
  - Research Site, Dortmund
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Geesthacht
  - Research Site, Gelsenkirchen
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Homburg
  - Research Site, Jena
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Magdeburg
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Neu-Isenburg
  - Research Site, Peine
  - Research Site, Potsdam
  - Research Site, Radebeul
  - Research Site, Reinfeld
  - Research Site, Rosenheim
  - Research Site, Schleswig
  - Research Site, Wiesbaden
  - Research Site, Witten
- Serbia (5):
  - Research Site, Belgrade
  - Research Site, Kamenitz
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Valjevo
- Slovakia (7):
  - Research Site, Bratislava
  - Research Site, Ilava
  - Research Site, Kežmarok
  - Research Site, Košice
  - Research Site, Poprad
  - Research Site, Prešov
  - Research Site, Žilina
- South Africa (20):
  - Research Site, Athlone
  - Research Site, Bellville
  - Research Site, Benoni
  - Research Site, Bloemfontein
  - Research Site, Boksburg
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, eMkhomazi
  - Research Site, Gatesville
  - Research Site, Johannesburg
  - Research Site, Kempton Park
  - Research Site, Kraaifontein
  - Research Site, Middelburg
  - Research Site, Mowbray
  - Research Site, Newtown
  - Research Site, Parktown
  - Research Site, Pretoria
  - Research Site, Roodepoort
  - Research Site, Umhlanga
  - Research Site, Witbank
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Madrid
  - Research Site, Mérida
  - Research Site, Valencia
- Ukraine (10):
  - Research Site, Cherkasy
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kherson
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya
- United Kingdom (16):
  - Research Site, Belfast
  - Research Site, Blackpool
  - Research Site, Bradford
  - Research Site, Chippenham
  - Research Site, Corby
  - Research Site, Kenilworth
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Newcastle upon Tyne
  - Research Site, Northwood
  - Research Site, Nottingham
  - Research Site, Peterborough
  - Research Site, Romford
  - Research Site, Shipley
  - Research Site, Sidcup
  - Research Site, Wokingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chipps BE, Albers FC, Reilly L, Johnsson E, Cappelletti C, Papi A. Efficacy and safety of as-needed albuterol/budesonide versus albuterol in adults and children aged >/=4 years with moderate-to-severe asthma: rationale and design of the randomised, double-blind, active-controlled MANDALA study. BMJ Open Respir Res. 2021 Dec;8(1):e001077. doi: 10.1136/bmjresp-2021-001077. PMID 34887317
- [Result] Papi A, Chipps BE, Beasley R, Panettieri RA Jr, Israel E, Cooper M, Dunsire L, Jeynes-Ellis A, Johnsson E, Rees R, Cappelletti C, Albers FC. Albuterol-Budesonide Fixed-Dose Combination Rescue Inhaler for Asthma. N Engl J Med. 2022 Jun 2;386(22):2071-2083. doi: 10.1056/NEJMoa2203163. Epub 2022 May 15. PMID 35569035
- [Derived] Chipps BE, Panettieri RA Jr, Skolnik N, Cappelletti C, Daoud SZ, Dunsire L, Gilbert IA, Papi A. Albuterol-budesonide rescue inhaler for asthma: Patterns of use and safety in the MANDALA trial. Ann Allergy Asthma Immunol. 2026 Jan;136(1):54-60.e3. doi: 10.1016/j.anai.2025.07.008. Epub 2025 Jul 13. PMID 40664332
- [Derived] Kew KM, Flemyng E, Quon BS, Leung C. Increased versus stable doses of inhaled corticosteroids for exacerbations of chronic asthma in adults and children. Cochrane Database Syst Rev. 2022 Sep 26;9(9):CD007524. doi: 10.1002/14651858.CD007524.pub5. PMID 36161875

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject enrolled on 13 December 2018 and the last subject completed the study on 07 February 2022. Subjects were enrolled at 347 study centers worldwide (Argentina, Canada, Czechia, Germany, Serbia, Slovakia, South Africa, Spain, Ukraine, United Kingdom and the United States).
Pre-assignment Details: The randomized treatment phase started after a 2 to 4 week screening period during which participants used sponsor provided Ventolin HFA (albuterol sulfate) as needed. In addition to the 3,132 participants randomized, 2,488 participants were screened but did not participate, of which 2,456 were ineligible (98.7%). The next most frequent reason was withdrawal by the participant, with 18 meeting this criteria.
Period: Overall Study
Arm/Group | BDA MDI (PT027) 160/180 μg | BDA MDI (PT027) 80/180 μg | AS MDI (PT007) 180 µg
Started | 1016 | 1057 | 1059
Completed | 915 | 933 | 916
Not Completed | 101 | 124 | 143
Not completed — Randomized and did not receive randomized study treatment | 1 | 2 | 2
Not completed — Withdrawal by Subject | 52 | 62 | 74
Not completed — Death | 4 | 2 | 2
Not completed — Adverse Event | 7 | 7 | 8
Not completed — A single severe exacerbation event lasting >20 days | 0 | 1 | 2
Not completed — >= 3 severe exacerbation events within a 3 month period | 1 | 4 | 4
Not completed — >= 5 total severe exacerbation events | 0 | 1 | 1
Not completed — Protocol Violation | 5 | 6 | 8
Not completed — Pregnancy | 1 | 0 | 3
Not completed — Lost to Follow-up | 19 | 25 | 21
Not completed — Condition under investigation worsened | 2 | 0 | 1
Not completed — Lack of Efficacy | 1 | 2 | 2
Not completed — Other reasons | 8 | 12 | 15

BASELINE CHARACTERISTICS:
Population: Of the 3,132 participants randomized, the full analysis set across all ages comprises 3,127 participants as one participant was randomized and did not receive randomized study treatment, and four participants were randomized in error and did not receive randomized study treatment. These five participants have therefore been excluded from the summaries of baseline characteristics, efficacy and safety.
Groups:
- Total: Total of all reporting groups
Arm/Group | BDA MDI (PT027) 160/180 μg | BDA MDI (PT027) 80/180 μg | AS MDI (PT007) 180 µg | Total
Number analyzed (Participants) | 1015 | 1055 | 1057 | 3127
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (15.05) | 48.5 (16.71) | 49.1 (17.22) | 49.4 (16.39)
Age, Customized [Count of Participants; unit: Participants]
  Children (>=4 to <12 years) | 0 | 41 | 42 | 83
  Adolescents (>=12 to <18 years) | 34 | 32 | 34 | 100
  Adults (>=18 to <65 years) | 789 | 805 | 784 | 2378
  Elderly (>=65 years) | 192 | 177 | 197 | 566
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 647 | 686 | 695 | 2028
  Male | 368 | 369 | 362 | 1099
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 235 | 261 | 316 | 812
  Not Hispanic or Latino | 780 | 794 | 741 | 2315
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 29 | 33 | 23 | 85
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 139 | 141 | 137 | 417
  White | 820 | 848 | 869 | 2537
  More than one race | 18 | 20 | 24 | 62
  Unknown or Not Reported | 8 | 12 | 4 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 19 | 11 | 12 | 42
  Argentina | 157 | 200 | 207 | 564
  United States | 274 | 275 | 290 | 839
  Czechia | 74 | 64 | 73 | 211
  Ukraine | 156 | 150 | 128 | 434
  South Africa | 106 | 120 | 115 | 341
  United Kingdom | 9 | 15 | 10 | 34
  Slovakia | 25 | 30 | 28 | 83
  Serbia | 65 | 54 | 57 | 176
  Germany | 109 | 108 | 112 | 329
  Spain | 21 | 28 | 25 | 74
Height [Mean (Standard Deviation); unit: Centimeters] | 166.8 (9.92) | 165.1 (11.45) | 164.4 (11.67) | 165.4 (11.10)
Weight [Mean (Standard Deviation); unit: Kilograms] | 80.5 (16.88) | 78.2 (18.93) | 78.8 (18.47) | 79.2 (18.15)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.887 (5.4002) | 28.496 (5.5886) | 28.948 (5.6271) | 28.776 (5.5432)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Severe Asthma Exacerbation Event
Description: Time to first severe asthma exacerbation will be calculated as the time from randomization until the start date of the first severe asthma exacerbation. An asthma exacerbation will be considered severe if it results in at least one of the following: a temporary bolus/burst of systemic corticosteroids for at least 3 consecutive days to treat symptoms of asthma worsening (a single depo-injectable dose of corticosteroids will be considered equivalent), an emergency room or urgent care visit (<24 hours in the facility for evaluation and treatment) due to asthma that required systemic corticosteroids, or an in-patient hospitalization (admission to an in-patient facility and/or ≥ 24 hours in a healthcare facility) due to asthma. The descriptive summary shows the number of participants with a severe exacerbation event, occurring between the date of randomization up to the date of randomized treatment discontinuation or a change in maintenance therapy.
Time Frame: From randomization up to a discontinuation of randomized treatment or a change in maintenance therapy. The mean and median reporting period for all participants was 44 and 48 weeks, respectively.
Population: All participants that were randomized, took at least one puff of randomized treatment, and had at least one efficacy assessment, excluding participants confirmed as duplicates (n = 4). As children <12 years of age were not randomized to the BDA MDI 160/180μg dose, comparison was made to the participants >=12 years of age within the AS MDI 180μg arm.
Measure: Count of Participants; unit: Participants
Groups:
- BDA MDI 160/180 μg (Full Analysis Set; >=12 Years): All participants who are randomized to BDA MDI 160/180 μg, are aged >=12 years at randomization, take at least one puff of randomized treatment and have at least one efficacy assessment, excluding participants identified as confirmed duplicates.
- AS MDI 180 μg (Full Analysis Set; >=12 Years): All participants who are randomized to AS MDI 180 μg, are aged >=12 years at randomization, take at least one puff of randomized treatment and have at least one efficacy assessment, excluding participants identified as confirmed duplicates.
- BDA MDI 80/180 μg (Full Analysis Set): All participants who are randomized to BDA MDI 80/180 μg, take at least one puff of randomized treatment and have at least one efficacy assessment, excluding participants identified as confirmed duplicates.
- AS MDI 180 μg (Full Analysis Set): All participants who are randomized to AS MDI 180 μg, take at least one puff of randomized treatment and have at least one efficacy assessment, excluding participants identified as confirmed duplicates.
Arm/Group | BDA MDI 160/180 μg (Full Analysis Set; >=12 Years) | AS MDI 180 μg (Full Analysis Set; >=12 Years) | BDA MDI 80/180 μg (Full Analysis Set) | AS MDI 180 μg (Full Analysis Set)
Number analyzed (Participants) | 1013 | 1014 | 1054 | 1056
Participants | 207 | 266 | 241 | 276
Statistical Analysis 1: Comparison: BDA MDI 160/180 μg (Full Analysis Set; >=12 Years) vs AS MDI 180 μg (Full Analysis Set; >=12 Years); H0 = null hypothesis. Hazard ratios, 95% confidence intervals for hazard ratios and p-values are estimated using a Cox regression model with treatment group, age group, region and number of severe exacerbations in the last 12 months prior to randomization as factors. A hazard ratio less than 1 favours BDA MDI treatment; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.733, 95% CI 2-sided [0.611 to 0.879]
Statistical Analysis 2: Comparison: BDA MDI 80/180 μg (Full Analysis Set) vs AS MDI 180 μg (Full Analysis Set); H0 = Null hypothesis. Hazard ratios, 95% confidence intervals for hazard ratios and p-values are estimated using a Cox regression model with treatment group, age group, region and number of severe exacerbations in the last 12 months prior to randomization as factors. A hazard ratio less than 1 favours BDI MDI treatment; Test type: Superiority; p = 0.041, Regression, Cox; Hazard Ratio (HR) = 0.835, 95% CI 2-sided [0.702 to 0.992]

2. Secondary Outcome: Annualized Severe Exacerbation Rate
Description: The annualized severe exacerbation rate (severe exacerbations per year) is estimated from a negative binomial model with treatment, age group, region, and number of severe exacerbations in the last 12 months prior to randomization as categorical covariates. The logarithm of the time at risk is included as an offset variable.
Time Frame: From randomization up to discontinuation of randomized treatment or a change in maintenance therapy. The mean and median reporting period for all participants was 44 and 48 weeks, respectively.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Severe exacerbations per year
Arm/Group | BDA MDI 160/180 μg (Full Analysis Set; >=12 Years) | AS MDI 180 μg (Full Analysis Set; >=12 Years) | BDA MDI 80/180 μg (Full Analysis Set) | AS MDI 180 μg (Full Analysis Set)
Number analyzed (Participants) | 1013 | 1014 | 1054 | 1056
Severe exacerbations per year | 0.45 [0.34 to 0.60] | 0.59 [0.44 to 0.78] | 0.49 [0.37 to 0.64] | 0.61 [0.46 to 0.80]
Statistical Analysis 1: Comparison: BDA MDI 160/180 μg (Full Analysis Set; >=12 Years) vs AS MDI 180 μg (Full Analysis Set; >=12 Years); Estimated from a negative binomial model with treatment, age group, region, and number of severe exacerbations in the last 12 months prior to randomization as categorical covariates. The logarithm of the time at risk is included as an offset variable. A sequential testing strategy is used for secondary endpoints. A null hypothesis can only be rejected if all preceding null hypotheses are also rejected; Test type: Superiority; p = 0.008, Negative binomial model; Rate Ratio = 0.76, 95% CI 2-sided [0.62 to 0.93]
Statistical Analysis 2: Comparison: BDA MDI 80/180 μg (Full Analysis Set) vs AS MDI 180 μg (Full Analysis Set); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.028, Negative binomial model; Rate Ratio = 0.8, 95% CI 2-sided [0.66 to 0.98]

3. Secondary Outcome: Total Annualized Dose of Systemic Corticosteroid (SCS)
Description: This endpoint includes all systemic corticosteroids (SCS) taken in response to a severe exacerbation event from randomization up to randomized treatment discontinuation or a change in maintenance therapy. All SCS are standardized to equipotent doses of prednisone before deriving the total dose. The total annualized dose is calculated as the total dose of SCS divided by the duration of the randomized treatment period.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Full Range); unit: Milligram(s)
Arm/Group | BDA MDI 160/180 μg (Full Analysis Set; >=12 Years) | AS MDI 180 μg (Full Analysis Set; >=12 Years) | BDA MDI 80/180 μg (Full Analysis Set) | AS MDI 180 μg (Full Analysis Set)
Number analyzed (Participants) | 1012 | 1011 | 1052 | 1052
Milligram(s) | 86.2 [0 to 3678] | 129.3 [0 to 18941] | 95.5 [0 to 4974] | 127.1 [0 to 18941]
Statistical Analysis 1: Comparison: BDA MDI 160/180 μg (Full Analysis Set; >=12 Years) vs AS MDI 180 μg (Full Analysis Set; >=12 Years); P-values are calculated via a Wilcoxon rank sum test. A sequential testing strategy is used for secondary endpoints. A null hypothesis can only be rejected if all preceding null hypotheses are also rejected; Test type: Superiority; p = 0.002, Wilcoxon rank sum
Statistical Analysis 2: Comparison: BDA MDI 80/180 μg (Full Analysis Set) vs AS MDI 180 μg (Full Analysis Set); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.06, Wilcoxon rank sum

4. Secondary Outcome: Asthma Control Questionnaire-5 (ACQ-5) - Number of Participants Who Were Responders at Week 24
Description: The ACQ-5 consists of 5 questions on symptom control, with each scored on a 7-point scale (0 = excellent asthma control; 6 = extremely poor control). The overall score (0 = excellent asthma control; 6 = extremely poor control, so a lower score is the better outcome) is the mean of the 5 symptom items. A responder is defined as a participant with a decrease from baseline to Week 24 overall ACQ-5 score of 0.5 or more. ACQ-5 is not validated for children less than 6 years old, data for participants who were 4 or 5 years old was excluded from the analysis of ACQ-5.
Time Frame: From baseline to Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BDA MDI 160/180 μg (Full Analysis Set; >=12 Years) | AS MDI 180 μg (Full Analysis Set; >=12 Years) | BDA MDI 80/180 μg (Full Analysis Set) | AS MDI 180 μg (Full Analysis Set)
Number analyzed (Participants) | 1013 | 1014 | 1052 | 1055
Participants | 677 | 630 | 681 | 650
Statistical Analysis 1: Comparison: BDA MDI 160/180 μg (Full Analysis Set; >=12 Years) vs AS MDI 180 μg (Full Analysis Set; >=12 Years); Logistic regression model with baseline ACQ-5 as a continuous covariate and age group, region and number of severe exacerbations in the 12 months prior to randomization as categorical covariates. A sequential testing strategy is used for secondary endpoints. A null hypothesis can only be rejected if all preceding null hypotheses are also rejected; Test type: Superiority; p = 0.033, Regression, Logistic; Odds Ratio (OR) = 1.221, 95% CI 2-sided [1.016 to 1.467]
Statistical Analysis 2: Comparison: BDA MDI 80/180 μg (Full Analysis Set) vs AS MDI 180 μg (Full Analysis Set); [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.175, Regression, Logistic; Odds Ratio (OR) = 1.132, 95% CI 2-sided [0.946 to 1.353]

5. Secondary Outcome: Asthma Quality of Life Questionnaire for Participants Aged 12 Years and Older (AQLQ+12) - Number of Participants Who Were Responders at Week 24
Description: The AQLQ+12 consists of 32 questions in 4 domains and is assessed on separate 7-point Likert scales from 1 to 7, with higher values indicating better health-related quality of life. The overall score is the mean of all responses. A responder is defined as a participant with an increase from baseline to week 24 AQLQ-12 score of at least 0.5.
Time Frame: From baseline to 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- BDA MDI 80/180 μg (Full Analysis Set; >=12 Years): All participants who are randomized to BDA MDI 80/180 μg, are aged >=12 years at randomization, take at least one puff of randomized treatment and have at least one efficacy assessment, excluding participants identified as confirmed duplicates.
Arm/Group | BDA MDI 160/180 μg (Full Analysis Set; >=12 Years) | BDA MDI 80/180 μg (Full Analysis Set; >=12 Years) | AS MDI 180 μg (Full Analysis Set; >=12 Years)
Number analyzed (Participants) | 994 | 987 | 993
Participants | 508 | 489 | 461
Statistical Analysis 1: Comparison: BDA MDI 160/180 μg (Full Analysis Set; >=12 Years) vs AS MDI 180 μg (Full Analysis Set; >=12 Years); Logistic regression model with baseline AQLQ-12 as a continuous covariate and age group, region and number of severe exacerbations in the 12 months prior to randomization as categorical covariates. A sequential testing strategy is used for secondary endpoints. A null hypothesis can only be rejected if all preceding null hypotheses are also rejected; Test type: Superiority; p = 0.028, Regression, Logistic; Odds Ratio (OR) = 1.228, 95% CI 2-sided [1.022 to 1.475]
Statistical Analysis 2: Comparison: BDA MDI 80/180 μg (Full Analysis Set; >=12 Years) vs AS MDI 180 μg (Full Analysis Set; >=12 Years); [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.26, Regression, Logistic; Odds Ratio (OR) = 1.111, 95% CI 2-sided [0.925 to 1.335]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time of signed informed consent/assent and up to the safety follow up period. Reported AEs are those that occurred from the date of first dose of randomized treatment up to the date of treatment discontinuation, which per protocol, was expected to be at least 24 weeks. The mean and median duration of exposure to randomized treatment for the reporting period for all participants was 44 and 48 weeks, respectively.
Arm/Group | BDA MDI (PT027) 160/180 μg | BDA MDI (PT027) 80/180 μg | AS MDI (PT007) 180 µg
All-Cause Mortality (participants affected / at risk) | 4/1015 | 2/1055 | 2/1057
Serious Adverse Events (participants affected / at risk) | 53/1015 | 40/1055 | 48/1057
Other Adverse Events (participants affected / at risk) | 244/1015 | 253/1055 | 243/1057
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BDA MDI (PT027) 160/180 μg (N=1015) | BDA MDI (PT027) 80/180 μg (N=1055) | AS MDI (PT007) 180 µg (N=1057)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 1 (3)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylatic shock (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Colpocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (9) | 20 (20)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 11 (12) | 5 (5) | 8 (8)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 4 (4) | 5 (5)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 4 (4) | 2 (2)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BDA MDI (PT027) 160/180 μg (N=1015) | BDA MDI (PT027) 80/180 μg (N=1055) | AS MDI (PT007) 180 µg (N=1057)
Hypertension (Vascular disorders) | 22 (23) | 27 (27) | 26 (27)
Headache (Nervous system disorders) | 44 (71) | 50 (77) | 49 (76)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (29) | 23 (23) | 20 (20)
Nasopharyngitis (Infections and infestations) | 76 (95) | 61 (68) | 54 (67)
COVID-19 (Infections and infestations) | 33 (33) | 47 (47) | 38 (38)
Upper respiratory tract infection (Infections and infestations) | 26 (31) | 31 (35) | 26 (28)
Bronchitis (Infections and infestations) | 25 (27) | 27 (30) | 28 (32)
Sinusitis (Infections and infestations) | 15 (16) | 17 (17) | 25 (28)
Influenza (Infections and infestations) | 21 (23) | 20 (22) | 14 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data or results obtained from this study must not be published without prior approval from the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT03769090/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT03769090/SAP_001.pdf